CLINICAL TRIAL: NCT02472925
Title: Way to Cure: Developing Effective Strategies to Promote Adherence to Hepatitis C Therapy Among Older Adults
Brief Title: Way to Cure HCV Adherence
Acronym: WTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P30AG034546 (NIH)
Record Dates: First submitted 2015-03-19; First posted 2015-06-16 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Control (Other): MedSignals pill box will be set into "quiet mode" to track patient compliance. This mode sends daily adherence data to the Way to Health platform each time the participant opens the pill box, however, does not remind the participant to take the medication.
  Interventions: Behavioral: MedSignals Pill Box
- Arm 2: Reminders/Feedback (Experimental): MedSignals pill box will track patient compliance and the Way to Health platform will allow participants to receive tailored text message reminders to take the medication if in case the interval from last cap opening is >30 hours (greater than 6 hours overdue).
  Interventions: Behavioral: MedSignals Pill Box
- Arm 3: Reminders/Feedback/Incentives (Experimental): MedSignals pill box will track patient compliance and in addition to reminders with missed doses and weekly adherence feedback, patients in this arm will be eligible to receive a small financial incentive each week they demonstrate perfect >85% adherence. The weekly adherence feedback message will also alert patients whether they earned the incentive for the past week.
  Interventions: Behavioral: MedSignals Pill Box

INTERVENTIONS:
Behavioral: MedSignals Pill Box — Pill box will provide feedback to the study team regarding subjects' compliance and provide reminders depending on Arm.

SUMMARY:
This is a 3-arm, multi-center, patient-randomized, field evaluation of the "Way to Cure" behavioral interventions on medication adherence in HCV.

DETAILED DESCRIPTION:
This 3-arm trial will field test the efficacy of "Way to Cure" intervention on medication adherence in Hepatitis C for 12 weeks. As part of routine clinical care all patients will receive medication counseling regarding proper use and side effects by trained nurses or pharmacists depending on the clinical site.

Arm 1: Control (n=20) - Monitoring pill box will be set into "quiet mode". This mode sends daily adherence data to the Way to Health platform each time the participant opens the pill bottle, however, does not remind the participant to take the medication. In the event no electronic signal is received by the platform for 96 hours, the RA will call the participant to assess any usability or connectivity issues.

Arm 2: Intervention - Reminders/Feedback (n=20) - Patients will receive tailored text message reminders to take the medication if in case the interval from last box opening is >30 hours (greater than 6 hours overdue). Patients will receive weekly text messages with summary cumulative adherence scores.

Arm 3: Intervention - Reminders/Feedback and Financial Incentives (n=20) - In addition to reminders with missed doses and weekly adherence feedback, patients in this arm will be eligible to receive a financial incentive each week they demonstrate perfect >85% adherence. The weekly adherence feedback message will also alert patients whether they earned the incentive for the past week.

ELIGIBILITY:
Inclusion Criteria:

a) age 50 older, b) prescribed a fixed dose combination HCV regimen containing sofosbuvir/ledipasvir for 12 weeks, and 3) willing to receive text message communications.

Exclusion Criteria:

a) non-English speaking, b) have severe vision, hearing impairment precluding study participation, c) no text messaging capability, d) decompensated cirrhosis requiring hospitalization in the past 30 days, e) medication primarily given by a caregiver/facility

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Pill bottle measured adherence | 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reese, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania